CLINICAL TRIAL: NCT00473304
Title: Contact Lens in Pediatrics (CLIP) in an Asian Population Study
Acronym: CLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: R501/50/2006
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia
Keywords: Safety; Efficacy; Adaptation; myopia and contact lens wear in children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Johnson&Johnson Acuevue daily disposable lenses

SUMMARY:
To evaluate the safety, efficacy and physiological performance of daily disposable spherical and toric soft contact lenses in a vision-corrected population of children ages 8-11 years of age. To evaluate the ability of the practitioner to fit these lenses and for the children to wear and manage these lenses.

DETAILED DESCRIPTION:
This is a bilateral, open-label dispensing evaluation of two daily lens types. Eligible subjects will wear the study lenses for 3-months daily wear. 1-Day Acuvue will be worn by spherical subjects and 1-Day Acuvue for Astigmatism will be worn by astigmats.

There is a total of 4 study visits (baseline, contact fitting and dispensing, 1 week, 1 month and 3 month follow-up). Tests conducted include manifest refraction and over-refraction, keratometry, visual acuity, ACA ratio, lens fit assessment, slit lamp biomicroscopy and parent/patient questionaires.

Each child was provided with a supply of lenses to last until the next scheduled follow-up visit, unit-dose rewetting drops for rinsing their lenses if necessary, and a daily log to complete each day until the next follow-up visit.

Informed consent was obtained from all subjects after the nature of the study had been fully explained. The study gained approval from the Ethics Committee of the Singapore Eye Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Be between 8-11 years of age.
* Signed Written Informed Consent and/or have the consent of a parent or legal guardian and Investigator to record this on Case Report Form (CRF) in appropriate space.
* Be a neophyte.
* Require a visual correction in both eyes.
* Require a soft contact lens spherical correction between +5.00 and -9.00 DS.
* Have an astigmatic correction between 0.00 amd 2.00 DC.
* Be able to wear the lens powers available for this study.
* Be correctable to a visual acuity of 20/25 or better in each eye.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  (i)No amblyopia. (ii) No evidence of lid abnormality or infection. (eg. entropion, ectropion, chalazia, recurrent styes). (iii) No clinically significant slit lamp (eg. any infiltrates or other slit lamp findings Grade 3 or above: corneal edema, corneal staining, tarsal abnormalities, conjunctival injection, vascularisation, or abnormal opacities).(iv) No other active ocular disease. (eg. glaucoma, history of recurrent corneal erosions, cornea infiltrates, conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology.)

Exclusion Criteria:

* Requires concurrent ocular medication.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* No clinically significant (Grade 3 or 4) slit lamp findings including corneal edema, corneal vascularization, corneal staining, tarsal abnormalities, bulbar injection, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Diabetic.
* Infectious disease (eg.hepatitis, tuberculosis)or an immunosuppressive disease (eg.HIV).
* PMMA or RGP lens wear in the previous 8 weeks.
* Has had refractive surgery. Has had eye injury/surgery within 8 weeks immediately prior to enrollment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrollment only.
* Participation in any concurrent clinical trial.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
i. demographics ii. refraction (D) visual acuity iii. AC/A Ratio (phorias in prism dioptres) iv. Keratometry v. Slit lamp examination vi. Corneal staining viii. Contact lens fit assessment | December 2006 to July 2007

SECONDARY OUTCOMES:
Questionaire filling by subject/parent | Dec 2006 to July 2007

CONTACTS AND LOCATIONS:
Overall Officials: Li Lim, FRCS(Ed), Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Sankaridurg PR, Sweeney DF, Holden BA, Naduvilath T, Velala I, Gora R, Krishnamachary M, Rao GN. Comparison of adverse events with daily disposable hydrogels and spectacle wear: results from a 12-month prospective clinical trial. Ophthalmology. 2003 Dec;110(12):2327-34. doi: 10.1016/S0161-6420(03)00795-4. PMID 14644714
- [Background] Suchecki JK, Ehlers WH, Donshik PC. A comparison of contact lens-related complications in various daily wear modalities. CLAO J. 2000 Oct;26(4):204-13. PMID 11071345
- [Background] Solomon OD, Freeman MI, Boshnick EL, Cannon WM, Dubow BW, Kame RT, Lanier JC Jr, Lopanik RW, Quinn TG, Rigel LE, Sherrill DD, Stiegmeier MJ, Teiche RS, Zigler LG, Mertz GW, Nason RJ. A 3-year prospective study of the clinical performance of daily disposable contact lenses compared with frequent replacement and conventional daily wear contact lenses. CLAO J. 1996 Oct;22(4):250-7. PMID 8906382